CLINICAL TRIAL: NCT03138759
Title: An Open-label, Randomized, 2-treatment, 2-period, Crossover Study to Evaluate the Effect of Probenecid on the Pharmacokinetics of Pexidartinib in Healthy Subjects
Brief Title: Effect of Probenecid on Pexidartinib Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PL3397-A-U122
Record Dates: First submitted 2017-04-28; First posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Pharmacokinetics in Healthy Volunteers
MeSH Terms: interventions — pexidartinib; Probenecid

STUDY DESIGN:
Intervention Model Description: This is an open-label, 2-treatment sequence, 2-period, crossover study with a washout between doses and treatment periods
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pexidartinib then Probenecid (Experimental): Participants receive Sequence AB: Treatment A (pexidartinib) first, then Treatment B (probenecid), with a washout period between them
  Interventions: Drug: Pexidartinib; Drug: Probenecid
- Probenecid then Pexidartinib (Experimental): Participants receive Sequence BA: Treatment B (probenecid) first, then Treatment A (pexidartinib), with a washout period between them
  Interventions: Drug: Pexidartinib; Drug: Probenecid

INTERVENTIONS:
Drug: Pexidartinib — Orally, on Day 2
  Other Names: Treatment A
Drug: Probenecid — Orally, on Day 2
  Other Names: Treatment B

SUMMARY:
The primary objective of this trial is to assess the effect of probenecid on the pharmacokinetics (PK) of single-dose pexidartinib in healthy subjects.

Secondary objectives are to assess the safety and tolerability of pexidartinib alone and in combination with probenecid.

Participants will be confined to the clinic for approximately 32 days. Blood samples will be collected for PK analysis of pexidartinib and metabolites at predose and up to 312 hours (h) post dose.

ELIGIBILITY:
Inclusion Criteria:

* Is a healthy, nonsmoking person with a body mass index of 18 kg/m2 to 30 kg/m2 (inclusive) at Screening
* Is willing to be confined at the clinic for approximately 32 days
* Is surgically sterile or a naturally postmenopausal female and not lactating, or a male who agrees to use double barrier methods of contraception and avoid donating sperm from Check-in until 90 d after the final dose of pexidartinib

Exclusion Criteria:

* Has any history or condition, per protocol or in the opinion of the investigator, that might compromise the participant's safety, their ability to complete the trial, and or analysis of results

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | predose to 312 hours post dose
  Maximum concentration of the drug and its metabolite in plasma
Time to Maximum Concentration (Tmax) | within 312 hours post dose
  Time at which the maximum concentration is reached
Area under the curve to the last quantifiable measurement (AUClast) | within 312 hours post dose
  Area under the drug concentration time curve from the first measurement to the last

SECONDARY OUTCOMES:
Number of participants experiencing an adverse event | within 312 hours post dose
  Total number of participants experiencing any adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo
Locations (1):
- Worldwide Clinical Trials Early Phase Services, San Antonio, Texas, United States

REFERENCES:
- [Derived] Zahir H, Greenberg J, Shuster D, Hsu C, Watanabe K, LaCreta F. Evaluation of Absorption and Metabolism-Based DDI Potential of Pexidartinib in Healthy Subjects. Clin Pharmacokinet. 2022 Nov;61(11):1623-1639. doi: 10.1007/s40262-022-01172-9. Epub 2022 Oct 20. PMID 36264536